CLINICAL TRIAL: NCT01750593
Title: Efficacy of Radiofrequency Ablation in Thyroid Nodules
Brief Title: Radiofrequency Ablation in Thyroid Nodules
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Yeliz Emine Ersoy, M.D., Bezmialem Vakif University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: yelizeminersoy
Record Dates: First submitted 2012-10-07; First posted 2012-12-17 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Thyroid Nodules
Keywords: radiofrequency; thyroid; nodule
MeSH Terms: conditions — Thyroid Nodule; Thyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- radiofrequency ablation of thyroid nodule (Experimental): Under ultrasonography the thyroid nodules will be ablated by radiofrequency ablation
  Interventions: Procedure: Radiofrequency ablation of the thyroid nodule

INTERVENTIONS:
Procedure: Radiofrequency ablation of the thyroid nodule — Under USG control, the nodule will be ablated by radiofrequency with a needle that has an active tip of 1 cm.

SUMMARY:
Thyroid nodules are common problems and although > 95% are stated to be benign, they may cause some problems like hyperthyroidism, compression symptoms, and cosmesis associated with their function, size and localization. Especially for these nodules, patients undergo surgery and face up with the problems associated with surgical complications although they are not cancer. In some studies, radiofrequency ablation previously used for intrabdominal tumors like hepatic metastasis...,was stated to be efficient in the treatment of benign thyroid nodules and in some recurrent thyroid cancer cases. Therefore, the investigators decided to use this method in our patients having nodules like previously mentioned and see the efficacy and safety of the technique.

ELIGIBILITY:
Inclusion Criteria:

1. the presence of subjective symptoms (foreign body sensation, neck discomfort or pain, compressive symptom) or cosmetic problems;
2. a poor surgical candidate or refusal to undergo surgery;
3. fine-needle aspiration cytology and US findings that were compatible with a benign nodule;
4. anxiety about a malignancy.

Exclusion Criteria:

1. a nodule less than 5 mm in size;
2. follicular neoplasm or malignancy on fine needle aspiration cytology (FNAC);
3. a nodule with the sonographic criteria for a malignancy (taller than wide, marked hypoechoic, microcalcifications, ill-defined margins), although FNAC was a benign result;
4. previous radiation or operation history to the head and neck; (5) previous sclerosing therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-01 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Shrinkage of the thyroid nodule after radiofrequency ablation | 6 months

SECONDARY OUTCOMES:
Disappearance of the nodules in follow up | 1 year

CONTACTS AND LOCATIONS:
Locations (3):
- Turkey (Türkiye) (3):
  - Bezmialem Vakif University, Istanbul, Istanbul
  - Bezmialem Vakif University medical Faculty, Istanbul
  - Bezmialem Vakif University, Istanbul